CLINICAL TRIAL: NCT05186649
Title: Left Atrial Appendage (LAA) Clot With Severe Mitral Stenosis, Responders and Non-responders With Anticoagulation
Brief Title: Left Atrial Appendage (LAA) Clot With Severe Mitral Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Karachi (Other)
Collaborators: Advanced Education & Research Center (Other); Karachi Institute of Heart Diseases (Network)
Responsible Party: Principal Investigator, Prof. Dr. Tariq Ashraf, Professor, University of Karachi
Other Study IDs: LAA-Pak-21
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Left Atrial Appendage Aneurysm; Mitral Stenosis
Keywords: Mitral Stenosis; Left Atrial Appendage; anticoagulation; echocardiography
MeSH Terms: conditions — Mitral Valve Stenosis | interventions — Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Group: Consecutive patients with severe mitral stenosis and clot in left atrial appendage (LAA) on transesophageal echocardiography fulfilling the inclusion criteria will be recruited for this study. An ACUSON 128-XP echocardiographic system equipped with omniplane and biplane transesophageal probes will be used for this study. TEE followed by CT Angiography will be performed according to the standard procedure after obtaining informed consent.
  Interventions: Other: WARFARIN

INTERVENTIONS:
Other: WARFARIN — 5 mg of daily dosage

SUMMARY:
Consecutive patients with severe mitral stenosis and clot in left atrial appendage (LAA) on transesophageal echocardiography fulfilling the inclusion criteria will be recruited for this study. An ACUSON 128-XP echocardiographic system equipped with omniplane and biplane transesophageal probes will be used for this study. TEE followed by CT Angiography will be performed according to the standard procedure after obtaining informed consent.

DETAILED DESCRIPTION:
Consecutive patients with severe mitral stenosis and clot in left atrial appendage (LAA) on transesophageal echocardiography fulfilling the inclusion criteria will be recruited for this study. An ACUSON 128-XP echocardiographic system equipped with omniplane and biplane transesophageal probes will be used for this study. TEE followed by CT Angiography will be performed according to the standard procedure after obtaining informed consent. Demographic profile of the patients will be recorded like gender and age. And baseline TEE will be interpreted and parameters such as mean MVO (cm2), mean MPG (mmHg), and mean LA size (AP diameter, cm) will be recorded. LAA morphologies will be classified as per the operational definition. All the patients will be put on oral anticoagulation with Warfarin. The international normalized ratio (INR) will be maintained between 2.5 and 3.5. Patients will be prescribed with warfarin initial with 5 mg of daily dosage. Weekly INR monitoring will be performed via weekly calls to each and every patients and their INR level will be obtained. Warfarin daily dosage will be adjusted after every month based on target INR range. Repeat TEE will be performed after three (3) months in all the patients. And presence and absence of clot in different types of LAA will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65 years.
* Both male and female.
* Patients with server mitral stenosis.
* Patients with LAA clot on TEE.
* Patients prescribed with anticoagulation (warfarin therapy).

Exclusion Criteria:

* Patients with severe MR
* Patients with severe AS
* Patients with NYHA class IV
* Patients whose valve morphology precluded PTMC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clot in left atrial appendage.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
frequency of left atrial appendage | 6 Month
  To determine frequency of left atrial appendage (LAA) clot resolution after three months of anticoagulation in patients with severe mitral stenosis.

SECONDARY OUTCOMES:
anatomies of LAA | 6 Month
  To assess the rate of response in different anatomies of LAA so that non-responders can be refer for surgery on the very first TEE examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Karachi Institute of Heart Disease, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Mahmood ul Hassan, Hussain C, Gul AM, ullah Jan H, Hafizullah M. Frequency of left atrial and appendage clot in patients with severe mitral stenosis. J Ayub Med Coll Abbottabad. 2010 Apr-Jun;22(2):40-2. PMID 21702263
- [Background] Mirdamadi A, Mirmohammadsadeghi M, Marashinia F, Nourbakhsh M. Left atrial appendage occlusion. Int J Prev Med. 2013 Jan;4(1):102-4. PMID 23411574
- [Background] Taghipour HR, Farahani MM, Ghiasi S, Naseri MH, Fakhraddin F. Coincidence of free-floating thrombus in the aortic arch, severe mitral stenosis, and left atrial appendage clot. Heart Surg Forum. 2011 Aug;14(4):E252-4. doi: 10.1532/HSF98.20101147. PMID 21859646
- [Background] Shibasaki I, Kaneko T, Obayashi T, Sato Y, Inaba H, Kaki N, Ogata T, Oki S. [A case of free-floating ball thrombus in left atrium with mitral stenosis]. Kyobu Geka. 2001 Mar;54(3):228-31. Japanese. PMID 11244757
- [Background] Oryoji A, Kawara T, Hara H, Aoyagi S, Kosuga K, Ohishi K. [Left atrial free-floating ball thrombus in a patient without mitral valve disease]. Nihon Kyobu Geka Gakkai Zasshi. 1993 Apr;41(4):699-703. Japanese. PMID 8515174
- [Background] Tremeau G, Chapon P, Buttard P, Gayet C, Oddou B, Nicolai Y, Beurlet J, Guichard G, Milon H. [Left atrial free floating thrombus without mitral valve disease. Review of the literature apropos of a case]. Arch Mal Coeur Vaiss. 1996 Jan;89(1):99-102. French. PMID 8678746